CLINICAL TRIAL: NCT02948361
Title: Clinical PRoduct DevelOpment StudyinG the QT Ultrasound® BReast ScannEr With Volunteer SubjectS
Acronym: PROGRESS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: QT Ultrasound LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR004
Record Dates: First submitted 2016-09-01; First posted 2016-10-28 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Volunteer Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QT Ultrasound breast scan (Experimental)
  Interventions: Other: QT Ultrasound Breast Scan

INTERVENTIONS:
Other: QT Ultrasound Breast Scan — Subjects will be scanned on the QT Ultrasound Breast Scanner. For subjects that may have breast calcifications and/or mass(es) and/or other finding(s) on the QT scan image(s), standard imaging modalities (e.g., mammogram and HHUS) will be performed per American College of Radiology (ACR) recommendations.

SUMMARY:
Subjects will be scanned on the QT Ultrasound Breast Scanner. For subjects that may have breast calcifications and/or mass(es) and/or other finding(s) on the QT scan image(s), standard imaging modalities (e.g., mammogram and HHUS) will be performed per ACR recommendations.

If available, subjects may provide copies of their breast imaging exams and related reports.

Demographics and medical history will be collected.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Willing and able to provide written, signed informed consent
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Inability to tolerate the scan
* Present infection risk
* Allergies to device materials
* Inability to successfully "fit" breast into the investigational device
* Currently pregnant as reported by the subject
* Body weight greater than 400 lbs. (180 kg)
* Any other conditions that the Investigator determines to interfere with the conduct of the study or evaluation of results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
QT Ultrasound scans | Scan session is 2 to 3 hours
  The capabilities of the QT Ultrasound scanner will be measured by the review of the QT Ultrasound scans at the conclusion of each QT Ultrasound scan session

CONTACTS AND LOCATIONS:
Locations (1):
- Marin Breast Health Trial Center, Novato, California, United States

IPD SHARING:
Plan to Share IPD: No